CLINICAL TRIAL: NCT01092858
Title: Effect of Exercise Alone or in Combination With Testosterone Replacement on Muscle Strength and Quality of Life in Older Men With Low Testosterone Concentrations: a Randomized Double-blind, Placebo Controlled Study
Brief Title: NEBIDO in Symptomatic Late Onset Hypogonadism (SLOH)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14853; 2009-017139-16 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Hypogonadism
Keywords: Testosterone undecanoate; Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate; testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Testosterone Undeconate (Nebido, BAY86-5037)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Undeconate (Nebido, BAY86-5037) — Testosterone undecanoate 1000 mg (4 ml) i.m. injection at baseline, at week 6, at week 18, at week 30 and at week 42, respectively
  Arms: Arm 1
Drug: Placebo — Matching placebo i.m. injections at baseline, at week 6, at week 18 at week 30 and at week 42, respectively
  Arms: Arm 2

SUMMARY:
The design of the study is a standard double-blind design, which is needed in this study to allow for unbiased evaluation of efficacy and safety. The effect of the additional impact of testosterone replacement therapy in hypogonadal men on muscle strength and quality of life in comparison to physical exercise alone will be assessed. Treatment duration will be 54 weeks, to monitor the increase as well as the "steady state" of the parameters assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 60 years and older (>60yrs), untrained
* Symptomatic hypogonadism as defined by a) and b)
* a) Total testosterone below 12 nmol/l (measurement 7.00-11.00 a.m.)
* b)Total Aging Males' symptom score above 36
* Willing to avoid significant change in the pattern of physical exercise and lifestyle for the duration of the study
* Residence in Cologne Area

Exclusion Criteria:

* Previous assignment to treatment during this study
* Use of androgen therapy or anabolic steroids respectively 12 months of entry into the study (i.e. screening visit/visit 1)
* Current participation in an exercise program or within the last 6 months
* Suspicion or known history of prostate or breast cancer or other hormone dependent neoplasia
* Abnormal finding on Digital Rectal Examination (DRE)
* Prostate specific antigen (PSA) level >4 ng/ml
* History of clinically significant post void residual urine (> 150 ml)
* Suspicion or known history of liver tumor
* Hypersensitivity to the active substances or any of the excipients of NEBIDO e.g. benzyl-benzoate and castor oil
* Blood coagulation irregularities presenting an increased risk of bleeding after intramuscular injections including vitamin-K-antagonists or other strong anticoagulants
* 32 Additional Exclusion Criteria

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Dynamic maximum strength -one repetition maximum (1-RM ) - of upper and lower extremity after 54 weeks | At baseline, at week 54

SECONDARY OUTCOMES:
Isometric maximum strength | At baseline, at week 54
Grip strength | At baseline, at week 54
Chair raising test | At baseline, at week 54
Arm curl test | At baseline, at week 54
Bicycle stress test with spirometry | At baseline, at week 54
SF-36 Questionnaire | At baseline, at week 54
AMS-Questionnaire | At baseline, at week 54
FINGER Questionnaire | At baseline, at week 54

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu